CLINICAL TRIAL: NCT05701462
Title: Role of B Mode and Color Doppler Sonography in Differentiation Between Pleural Neoplasm and Inflammatory Pleural Thickening in Correlation With CT Findings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Harby Mohamed, resident at diagnostic radiology department at Sohag general hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-01-04
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Pleural Thickening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pleural disease (Experimental)
  Interventions: Diagnostic Test: biopsy under sonographic gidance

INTERVENTIONS:
Diagnostic Test: biopsy under sonographic gidance — pleural biopsy under sonographic guidance

SUMMARY:
pleura is a serous membrane, it consist of parietal pleura and visceral pleura. pleural thickening is any form of thickening involving the pleura more than 3 mm.

there is malignant thickening : methoselioma, metastasis and non malignant thickening.

trans thoracic USn is a reliable , safe and gold standard for studying pleura.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed as having pleural thickening with or without pleural effusion.

Exclusion Criteria:

* Emphysema or contraindication to pleural biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity of sonography in pleural thickening in comparison to CT and histopathology | one year
  sensitivity of sonography in cases of pleural thickening in comparison to CT findings and histopathology

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Porcel JM. Pleural ultrasound for clinicians. Rev Clin Esp (Barc). 2016 Nov;216(8):427-435. doi: 10.1016/j.rce.2016.05.009. Epub 2016 Jun 6. English, Spanish. PMID 27282205
- [Background] Hallifax RJ, Haris M, Corcoran JP, Leyakathalikhan S, Brown E, Srikantharaja D, Manuel A, Gleeson FV, Munavvar M, Rahman NM. Role of CT in assessing pleural malignancy prior to thoracoscopy. Thorax. 2015 Feb;70(2):192-3. doi: 10.1136/thoraxjnl-2014-206054. Epub 2014 Jul 30. PMID 25077699
- [Background] Sureka B, Thukral BB, Mittal MK, Mittal A, Sinha M. Radiological review of pleural tumors. Indian J Radiol Imaging. 2013 Oct;23(4):313-20. doi: 10.4103/0971-3026.125577. PMID 24604935
- [Background] Pairon JC, Laurent F, Rinaldo M, Clin B, Andujar P, Ameille J, Brochard P, Chammings S, Ferretti G, Galateau-Salle F, Gislard A, Letourneux M, Luc A, Schorle E, Paris C. Pleural plaques and the risk of pleural mesothelioma. J Natl Cancer Inst. 2013 Feb 20;105(4):293-301. doi: 10.1093/jnci/djs513. Epub 2013 Jan 25. PMID 23355760